CLINICAL TRIAL: NCT04659421
Title: A Prospective, Singal-arm Clinical Study of Recombinant Human Endostatin (ENDOSTAR) Combined With Carboplatin and Vincristine in the Treatment of Low-grade Gliomas in Children
Brief Title: Study of Recombinant Human Endostatin Combined With CV Regimen in the Treatment of Pediatric Low-grade Gliomas
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Beijing Sanbo Brain Hospital (Other)
Responsible Party: Principal Investigator, Junping Zhang, Chief physician, Beijing Sanbo Brain Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SBNK-YJ-2020-016-02
Record Dates: First submitted 2020-11-24; First posted 2020-12-09 (Actual); Last update posted 2023-07-24 (Actual); Status verified 2023-07

CONDITIONS: Low-grade Glioma; Pediatric Brain Tumor
MeSH Terms: interventions — Psychotherapy, Multiple

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Low-grade gliomas (Experimental): Treated with Recombinant human endostatin, Carboplatin, and Vincristine
  Interventions: Drug: combined therapy with rh-ES and CV

INTERVENTIONS:
Drug: combined therapy with rh-ES and CV — All the patients receive combined therapy with recombinant human endostatin and traditional weekly CV regimen.
  Carboplatin is administered at a dose of 220 mg/m2. Vincristine is administered at a dose of 1.5 mg/m2 (maximum dose 2 mg). Recombinant human endostatin (rh-ES) is administrated at a dose of 15mg daily, for 14 consecutive days every 3 weeks.

SUMMARY:
Low-grade gliomas (LGGs) are the most common intracranial tumors in children, accounting for about 40% of intracranial tumors in children. The biological characteristics and clinical prognosis of LGGs vary greatly, and they can present different biological characteristics such as restricted growth, invasive growth, and malignant transformation during their development. The prognosis of LGGs is related to the degree of tumor resection, histological type, and whether it has spread.

For LGGs, surgical resection is the main treatment method. However, many tumors located in the visual pathway, brainstem, hypothalamus and other midline parts, it is impossible to completely remove. Radiotherapy can effectively control tumor progression to a certain extent, but radiotherapy can cause obvious and serious delayed damage, such as cognitive impairment, endocrine disorders, cerebrovascular events, and second tumors. Chemotherapy can effectively treat LGGs in children, and can postpone or avoid radiotherapy. It is the preferred treatment for children with LGGs after surgery. Carboplatin combined with vincristine, the CV regimen, is currently the main chemotherapy regimen for the treatment of children with LGGs.

Anti-angiogenesis is a new type of treatment. Bevacizumab, a humanized monoclonal antibody that targets vascular endothelial growth factor (VEGF). Among children with relapsed, refractory or progressing LGGs, the effective rate of Bev combined with irinotecan was 44%, and the 6-month and 2-year progression-free survival rates were 85% and 48%, respectively. However, almost all of them were treated with Bev progressed again. Tumor growth is more aggressive after Bev treatment fails. Recombinant human endostatin (rh-ES) is an endogenous broad-spectrum angiogenesis inhibitor that has been shown to significantly improve therapeutic efficacy when combining with conventional chemotherapy agents in non-small-cell lung cancer, breast cancer and melanoma.Previous retrospective studies of the research team found that rh-ES combined with CV can treat LGGs in children effectively, shorten the onset time, help quickly alleviate the symptoms of brainstem damage, and improve the quality of life.

This study intends to use prospective clinical studies to further confirm the efficacy and safety of the anti-angiogenic drug rh-ES combined with traditional CV regimens in the treatment of children with LGGs.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 3months and ≤18years;
2. Histopathologically confirmed low-grade glioma (WHO grade I and II), including astrocytoma, pilocytic astrocytoma, pleomorphic xanthoastrocytoma, subependymal giant cell astrocytoma, infantile desmoplastic astrocytoma, low-grade oligodendroglioma, oligoastrocytoma, ganglioglioma, and infantile desmoplastic ganglioglioma. Chiasmatic-hypothalamic tumors intrinsic to the optic pathway were eligible without pathologic confirmation.
3. There is a clear evaluable lesion with less than 95% resection or residual tumor of more than 1.5 cm^2；
4. KPS score ≥50 (age> 12 years old) or Lansky score ≥ 50 (age ≤ 12 years old)；
5. Estimated survival of at least 12 weeks;
6. Have not been received radiotherapy or chemotherapy before；
7. Participants must have adequate organ function as defined by the following criteria (within 7 days before treatment):

   Hematology (No transfusion within 14 days):

   Hemoglobin(HB)≥90g/L; Absolute neutrophil count (ANC)≥1.5×10^9/L; Platelet (PLT)≥80×10^9/L.

   Chemistry:

   Serum bilirubin ≤ 1.5×upper limit of normal (ULN) ALT and AST≤2.5ULN； Serum creatinine ≤1.5ULN or creatinine clearance rate(CCr)≥60ml/min； ECG: heart rate in the normal range (55-100beats/min), normal or slightly prolonged QT interval (QTc<480ms), normal or low T wave, normal or non-specific ST segment changes；
8. The patient or his legal guardian signs an informed consent form.

Exclusion Criteria:

1. MRI examination is not available;
2. Diffuse intrinsic pontine glioma or diffuse midline glioma with H3K27 mutation, even though the histopathology is grade I/II;
3. Non-glial low-grade rare intracranial tumors;
4. Receiving any other investigational agent;
5. History of allergic reactions attributed to compounds of similar chemical or biologic composition to the drugs used in this study;
6. Patients who have received organ transplants;
7. Patients with HIV or Treponema pallidum infection;
8. Severe heart disease; ECG shows T wave inversion or elevation or ST segment specific changes;
9. There were clinically significant bleeding symptoms or clear bleeding tendency in the first 3 months before enrollment, such as gastrointestinal bleeding, hemorrhagic gastric ulcer, gastrointestinal perforation, baseline fecal occult blood ++ and above, intracranial or intracranial hemorrhage, or vasculitis;
10. Arteriovenous thrombosis events occurred within 6 months before enrollment, such as cerebrovascular accidents (including temporary ischemic attack, cerebral hemorrhage, cerebral infarction), deep vein thrombosis and pulmonary embolism, etc.;
11. Having bleeding disorder and are being treated with thrombolytic or anticoagulant drugs.
12. Patients who are pregnant or breastfeeding.
13. Other conditions considered inappropriate by the researcher for inclusion.

Ages: 3 Months to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 60 (Actual)
Dates: Start 2020-11-03 (Actual); Primary Completion 2023-07-01 (Actual); Study Completion 2023-07-20 (Actual)

PRIMARY OUTCOMES:
objective response rate | up to 5years
  the percentage of patients who achieved confirmed complete response or partial response according to the Response Assessment in Neuro-Oncology (RANO) criteria

SECONDARY OUTCOMES:
median time to response | up to 5years
  Time interval from the beginning of chemotherapy to achieving CR, PR or MR
Progression-free survival | up to 5years
  the time interval from treatment initiation to disease progression or death, whichever occurs first.
Overall survival | up to 5years
  the time interval from treatment initiation to death from any cause.
The correlation between KPS change and efficacy | up to 5years
  the correlation between KPS baseline, KPS change (increase, decrease,stable) and best efficacy (CR, PR, SD, PD).
Frequency and severity of treatment-related adverse events as assessed by CTCAE v5.0 | up to 5years
  Frequency and severity of treatment-related adverse events as assessed by Common Terminology Criteria for Adverse Events (CTCAE) version 5.0

CONTACTS AND LOCATIONS:
Locations (1):
- Capital Medical University Sanbo Brain Hospital, Beijing, China